CLINICAL TRIAL: NCT03476889
Title: A Randomised, Controlled, Double-blind, Parallel Group, Multi-country Study to Investigate the Safety and Tolerance of a Partly Fermented Infant Formula Containing Prebiotic Oligosaccharides in Healthy Term Infants
Brief Title: Safety and Tolerance of a Partly Fermented Infant Formula With Prebiotic Oligosaccharides in Healthy Infants
Acronym: VOYAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EBB17TA14644
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-03

CONDITIONS: Growth
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Cows milk based infant formula containing fermented infant formula and prebiotic oligosaccharides
  Interventions: Other: Infant formula
- Control (Active Comparator): Cows milk based infant formula containing prebiotic oligosaccharides (commercially available Aptamil ProNutra)
  Interventions: Other: Infant formula
- Breastfed reference (No Intervention): Exclusively breastfed from birth to study completion

INTERVENTIONS:
Other: Infant formula — Infants are randomized to one of two infant formulas from <14 days of age to 17 weeks of age.
  Arms: Control; Intervention

SUMMARY:
A randomised, controlled, double-blind, parallel group, multi-country study to investigate the safety and tolerance of a partly fermented infant formula containing prebiotic oligosaccharides in healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, singleton, term infants
2. Aged ≤14 days at randomisation/enrolment
3. Birth weight within normal range for gestational age and sex
4. Head circumference at birth within normal range for age and sex
5. Maternal age ≥18 years at birth;
6. Intervention arms: exclusively formula fed at randomisation (infants of mothers who autonomously chose not to breastfeed for any reason before their infant is ≤14 days of age, and who intend to exclusively formula feed until their infant is at least 17 weeks of age); OR Breastfed reference arm: exclusively breastfed at enrolment (infants of mothers who intend to exclusively breastfeed until their infant is at least 17 weeks of age);
7. Written informed consent from parent(s) and/or legal guardian(s), who themselves are aged ≥18 years.

Exclusion Criteria:

1. Infants who require to be fed a special diet other than standard cow's milk based infant formula;
2. Infants known or suspected to have cow's milk allergy, soy allergy and/or lactose intolerance;
3. Infants known or suspected to have current or previous illnesses/conditions or interventions which could interfere with the study or its outcome parameters, as per the clinical judgement of the Investigator;
4. Infants with known or suspected congenital diseases or malformations which could interfere with the study or its outcome parameters (including, but not limited to: GI malformations, congenital immunodeficiency), as per the clinical judgement of the Investigator;
5. Infants with previous, current or intended participation in any other clinical study involving investigational or marketed products;
6. Incapability of infants' parents/legally acceptable representatives to comply with study protocol or Investigator's uncertainty about the willingness or ability of the parent(s)/legally acceptable representative(s) to comply with the protocol requirements;
7. Infants born from mothers with significant medical conditions during pregnancy that might interfere with the study or known to affect intra-uterine growth (e.g. placenta previa, pre-eclampsia, eclampsia, gestational diabetes requiring insulin or oral medication) as per Investigator's judgement.

   Criteria for lactating mothers of subjects in the breastfed reference arm:
8. Lactating women who are currently participating or intend to participate in any other clinical study involving investigational products. Participation in purely observational studies is permitted;
9. Lactating women known to suffer from hepatitis B or human immunodeficiency virus;
10. Lactating women known to have any other significant medical condition(s) which might interfere with the study or its outcome parameters (breast abscess or mastitis which could interfere with lactation, or other clinically relevant infections, or consumption of medication/substances which could impact the infants' growth), as per the clinical judgement of the Investigator;
11. Lactating women who intend to feed their infants with a combination of human milk and infant formula.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Weight gain (infant formula comparison) | 17 weeks
  Equivalence of weight gain per day (g/d) from baseline until 17 weeks of age in subjects receiving the test product compared to infants receiving the control product

SECONDARY OUTCOMES:
Weight gain (human milk comparison) | 17 weeks
  Equivalence of weight gain per day (g/d) from baseline until 17 weeks of age in subjects receiving the test product compared to infants receiving human milk
Recumbent Length gain | 17 weeks
  Equivalence of length gain per day (mm/d) from baseline until 17 weeks of age in subjects receiving the test product compared to infants receiving the control product or human milk
Head circumference gain | 17 weeks
  Equivalence of head circumference gain per day (mm/d) from baseline until 17 weeks of age in subjects receiving the test product compared to infants receiving the control product or human milk
Parent-reported GI Tolerance Parameters (daily diary) | 17 weeks
  Information on regurgitation and vomiting will be collected by a daily diary that is completed by the parents.
Parent-Reported Stool Characteristics (adapted Amsterdam Stool Scale) | 17 weeks
  Information on stool consistency (4-point scale) and stool frequency (number of stools per day) will be collected by a daily diary that is completed by the parents. Occurrence of diarrhea like-symptoms and constipation-like symptoms will be derived from the stool frequency and consistency data.
Incidence of treatment-related adverse events | 17 weeks
  Number of adverse events (by "System/Organ Class" and "Preferred term" according the MedDRA) as assessed and reported by the investigator.
Severity of treatment-related adverse events | 17 weeks
  Severity of adverse events (by "System/Organ Class" and "Preferred term" according the MedDRA) as assessed and reported by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinika Ginekologiczno-Położnicza Sp. z o.o. Sp. k., Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Undecided